CLINICAL TRIAL: NCT06193148
Title: A Study to Evaluate the Effect of Oral Administration of Jaktinib Hydrochloride Tablets on QT/Corrected QT (QTc) Interval in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Jaktinib on QT/QTc Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZGJAK039
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Jaktinib 100mg (Experimental): 6 Participants will receive Jaktinib 100 mg, orally; 2 Participants will receive placebo, orally.
  Interventions: Drug: Jaktinib; Drug: Placebo
- Jaktinib 400mg (Experimental): 6 Participants will receive Jaktinib 400 mg, orally; 2 Participants will receive placebo, orally.
  Interventions: Drug: Jaktinib; Drug: Placebo
- Jaktinib 600mg (Experimental): 6 Participants will receive Jaktinib 600 mg, orally; 2 Participants will receive placebo, orally.
  Interventions: Drug: Jaktinib; Drug: Placebo
- Jaktinib 800mg (Experimental): 6 Participants will receive Jaktinib 800 mg, orally; 2 Participants will receive placebo, orally.
  Interventions: Drug: Jaktinib; Drug: Placebo

INTERVENTIONS:
Drug: Jaktinib — Participants will receive Jaktinib orally for single dose
Drug: Placebo — Participants will receive Placebo orally for single dose

SUMMARY:
To evaluate the effect of Jaktinib Hydrochloride Tablets on QT/QTc interval in healthy subjects after a single oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent, able to comply with the requirements of the study.
* Age 18-45 years old, both male and female;
* Weight: male ≥ 50 kg, female ≥ 45 kg, 19 kg/m^2 ≤ BMI ≤26 kg/m^2.
* 12-lead electrocardiogram (ECG) examination, 300 ms≤QTcF<450 ms, 120 ms≤PR interval ≤200 ms, and QRS duration <120 ms;
* The subjects (including male subjects) are willing to voluntarily take effective contraceptive measures within the next 3 months.

Exclusion Criteria:

* Have a history of risk factors for torsade de pointes, or have a family history of short QT syndrome, long QT syndrome, unexplained sudden death in young adulthood (≤40 years old), drowning or sudden infant death syndrome in first-degree relatives;
* Previous history of hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia;
* Subjects who had donated blood or lost ≥400 mL of blood within 3 months before screening;
* HBsAg, HCV antibody, HIV antibody, or TP antibody antibody positive.
* Women with positive blood pregnancy test (applicable to women) or lactating women;
* Subjects who have other factors that the investigator considers unsuitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
QT Interval Corrected Using Fridericia's Formula | From before dosing until 48 hours after dosing
  Model-guided placebo-corrected change in QTcF from baseline (ΔΔQTcF)

CONTACTS AND LOCATIONS:
Overall Officials: LiYan Miao, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhu, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided